CLINICAL TRIAL: NCT00361894
Title: RECORD 3 Study: REgulation of Coagulation in ORthopedic Surgery to Prevent DVT and PE; a Controlled., Double-blind, Randomized Study of BAY 59-7939 in the Prevention of VTE in Subjects Undergoing Elective Total Knee Replacement.
Brief Title: Regulation of Coagulation in Orthopedic Surgery to Prevent Deep Vein Thrombosis (DVT) and Pulmonary Embolism (PE). A Study of BAY 59-7939 in the Prevention of VTE in Subjects Undergoing Elective Total Knee Replacement.
Acronym: RECORD 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11356; EudraCT: 2005-004620-40
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Prevention; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 2 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — 10 mg rivaroxaban (tablet) once daily administered for 13 +/- 2 days
  Arms: Arm 1
Drug: Enoxaparin — Syringe of enoxaparin at a dose of 40 mg for 13 +/- 2 days
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if 10 mg Bay 59-7939, taken once daily as a tablet, is safe and prevents blood clot which may form after a knee replacement operation.

ELIGIBILITY:
Inclusion Criteria:- Male and female patients aged 18 years or above- Patients scheduled for elective total knee replacement Exclusion Criteria:- Active bleeding or high risk of bleeding contraindicating treatment with LMWH- Contraindication listed in the labeling or conditions precluding subject treatment with enoxaparin or requiring dose adjustment (e.g. severe renal impairment, please refer to the local label of enoxaparin in your country)- Conditions prohibiting bilateral venography (e.g. amputation of 1 leg, allergy to contrast media)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2531 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of total VTE i.e.: Any DVT (proximal and/or distal), Non fatal PE, Death of all causes | Treatment period: up to Day 13+/-4

SECONDARY OUTCOMES:
Incidence of the composite endpoint comprising proximal DVT, non-fatal PE and VTE- related death (major VTE) | Treatment period: up to Day 13+/-4
Incidence of symptomatic VTE (DVT, PE) | Treatment period: up to Day 13+/-4
Incidence of DVT (total, proximal, distal) | Treatment period: up to Day 13+/-4
Incidence of symptomatic VTE during follow-up | Follow-up period: following 13+/-4 days
The composite endpoint comprising major VTE and treatment-emergent major bleeding | For major VTE, treatment period: up to Day 13+/-4 ; for major bleeding, from first dose of double-blind study medication to up to two days after last dose of double-blind study medication
Incidence of the composite endpoint that results from the primary endpoint by substituting VTE related death for all death | Treatment period: up to Day 13+/-4
Incidence of the composite endpoint that results from major VTE by substituting all cause mortality for VTE-related death | Treatment period: up to Day 13+/-4
Treatment-emergent major bleedings | From first dose of double-blind study medication to up to two days after last dose of double-blind study medication

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (127):
- Austria (4):
  - Graz, Styria
  - Innsbruck, Tyrol
  - Linz, Upper Austria
  - Vienna, Vienna
- Belgium (7):
  - Antwerp
  - Hasselt
  - Liège
  - Merksem
  - Pellenberg
  - Reet
  - Roeselare
- Canada (10):
  - Penticton, British Columbia
  - Saint John, New Brunswick
  - Burlington, Ontario
  - Kitchener, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Scarborough Village, Ontario
  - Windsor, Ontario
- China (2):
  - Beijing
  - Shanghai
- Colombia (3):
  - Bogotá
  - Cali
  - Medellín
- Czechia (8):
  - Prague, Tschechien
  - Brno
  - Chomutov
  - Havlíčkův Brod
  - Jihlava
  - Kolín
  - Pardubice
  - Pilsen
- Denmark (5):
  - Frederiksberg
  - Hellerup
  - Herlev
  - Hørsholm
  - Silkeborg
- France (10):
  - Bois-Guillaume
  - Clermont-Ferrand
  - Liévin
  - Marseille
  - Monaco
  - Nantes
  - Nice
  - Paris
  - Soyaux
  - Vandœuvre-lès-Nancy
- Germany (10):
  - Bad Mergentheim, Baden-Wurttemberg
  - Rheinfelden, Baden-Wurttemberg
  - Fürth, Bavaria
  - Garmisch-Partenkirchen, Bavaria
  - Würzburg, Bavaria
  - Sommerfeld, Brandenburg
  - Bremen, City state Bremen
  - Frankfurt am Main, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
- Israel (7):
  - Beersheba, Israel
  - Haifa, Israel
  - Holon, Israel
  - Kfar Saba, Israel
  - Tel Aviv, Israel
  - Ẕerifin, Israel
  - Tel Litwinsky
- Italy (12):
  - San Donato Milanese, Milano
  - Abano Terme, Padova
  - Gubbio, Perugia
  - Alghero, Sassari
  - Bologna
  - Florence
  - Lecco
  - Padua
  - Parma
  - Roma
  - Udine
  - Varese
- Mexico (3):
  - Chihuahua, Chih., Chihuahua
  - Guadalajara, Jalisco
  - Hermosillo, Sonora
- Netherlands (7):
  - Amsterdam
  - Hilversum
  - Hoofddorp
  - Leiden
  - Nijmegen
  - Oss
  - Zwolle
- Norway (5):
  - Elverum
  - Gjøvik
  - Kongsvinger
  - Lillehammer
  - Namsos
- Peru (2):
  - Callao
  - Lima
- Poland (8):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Szczecin
  - Warsaw
- South Africa (8):
  - Bloemfontein, Freestate
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Randburg, Gauteng
  - Durban, KwaZulu-Natal
  - Newcastle, KwaZulu-Natal
  - Somerset West, Western Cape
  - Worcester, Western Cape
- Spain (8):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Castellon, Castellón de La Plana
  - Jaén, Jaén
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Pamplona, Pamplona
  - Valencia, Valencia
- Sweden (8):
  - Falköping
  - Gothenburg
  - Halmstad
  - Hässleholm
  - Jönköping
  - Kungälv
  - Lidköping
  - Varberg

REFERENCES:
- [Derived] Lassen MR, Ageno W, Borris LC, Lieberman JR, Rosencher N, Bandel TJ, Misselwitz F, Turpie AG; RECORD3 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty. N Engl J Med. 2008 Jun 26;358(26):2776-86. doi: 10.1056/NEJMoa076016. PMID 18579812
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/